CLINICAL TRIAL: NCT02291120
Title: MEDCEM PC and MTA in Pulpotomies of Primary Molars
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Cristina Cuadros, Master's Program Director in Pediatric Dentistry, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIC-ODP-4
Record Dates: First submitted 2014-06-27; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Evaluate the Effects of MEDCEM PC and MTA in Pulpotomies of Primary Molars.
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- MTA (Active Comparator): ProRoot® MTA is a root canal repair material that is a unique improvement over other materials used for root canal repair. Made up of fine hydrophilic particles that set in the presence of water, ProRoot® MTA seals off all pathways between the root canal system and surrounding tissues, significantly reducing bacterial migration. Its excellent compatibility with the dentinal wall allows for a predictable clinical healing response.
  Interventions: Procedure: Pulpotomy
- MedCem Portland Cement (PC) (Experimental): MedCem PC is an excellent capping material for cariology on permanent teeth (direct and indirect capping) and in milk tooth endodontics (milk tooth amputation). Is characterized by excellent colour stability and neutrality and does not contain any additional ingredients
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy

SUMMARY:
The objective of the study is to evaluate and compare, clinically and radiographically,the effects of MEDCEM PC and MTA when used as pulp dressings following pulpotomy in human primary molars.

ELIGIBILITY:
Inclusion Criteria:

* healthy children
* molars showing: symptomless exposure of vital pulp by caries no clinical or radiographic evidence of pulp degeneration (excessive bleeding from the root canal, internal root resorption, inter-radicular and/or furcal bone destruction) the possibility of proper restoration of the teeth no physiological resorption of more than one-third of the root

Exclusion Criteria:

* presence of systemic pathology
* history of allergic reaction to latex, local anaesthetics or to the constituents of the test pulp dressing agents

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 24 months
  No pain, no swelling, no fistula or sinus tract, no pathologic mobility
Radiographic success | 24 months
  No internal root resorption progressing into the bone, no external root resorption, no furcation and/or periapical bone destruction

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain